CLINICAL TRIAL: NCT06340308
Title: Clinical Study With Berberine-based Food Supplement, Artichoke Extract, Phytosterols, Fenugreek and SelectSIEVE® OptiChol
Acronym: PARAF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PARAF 986117570
Record Dates: First submitted 2024-03-23; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Phytosterols; fenugreek seed meal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 tablet (Experimental)
  Interventions: Dietary Supplement: Berberine-based Food Supplement, Artichoke Extract, Phytosterols, Fenugreek and SelectSIEVE® OptiChol
- 2 tablets (Active Comparator)
  Interventions: Dietary Supplement: Berberine-based Food Supplement, Artichoke Extract, Phytosterols, Fenugreek and SelectSIEVE® OptiChol

INTERVENTIONS:
Dietary Supplement: Berberine-based Food Supplement, Artichoke Extract, Phytosterols, Fenugreek and SelectSIEVE® OptiChol — Patients will take 1 tablet of Berberine-based Food Supplement, Artichoke Extract, Phytosterols, Fenugreek and SelectSIEVE® OptiChol for 12 weeks
  Arms: 1 tablet
Dietary Supplement: Berberine-based Food Supplement, Artichoke Extract, Phytosterols, Fenugreek and SelectSIEVE® OptiChol — Patients will take 2 tablets of Berberine-based Food Supplement, Artichoke Extract, Phytosterols, Fenugreek and SelectSIEVE® OptiChol for 12 weeks
  Arms: 2 tablets

SUMMARY:
To evaluate the effects of a nutraceutical containing Berberine-based Food Supplement, Artichoke Extract, Phytosterols, Fenugreek and SelectSIEVE® OptiChol on lipid profile

DETAILED DESCRIPTION:
To evaluate the effects of a nutraceutical containing Berberine-based Food Supplement, Artichoke Extract, Phytosterols, Fenugreek and SelectSIEVE® OptiChol compared to placebo on lipid profile in patients with LDL cholesterol > 115 and < 190 mg/dl.Patients were allocated to receive 1 or 2 tablets of the nutraceutical for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* LDL Cholesterol > 115 mg/dl and < 190 mg/dl
* primary prevention

Exclusion Criteria:

* patients with neoplastic and liver diseases, renal failure and diabetes mellitus
* pregnant or breastfeeding women
* hypersensitivity to any of the ingredients
* therapy with lipid-lowering drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Variations of lipid profile | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico S. Matteo Foundation, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No